CLINICAL TRIAL: NCT04671771
Title: A Study to Evaluate the Safety and Effectiveness of the InnAVasc Arteriovenous Graft for Hemodialysis Access in Patients With End-Stage Renal Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: W.L.Gore & Associates (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSP-2002
Record Dates: First submitted 2020-12-05; First posted 2020-12-17 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: End Stage Renal Disease (ESRD); Kidney Failure; Chronic Renal Disease; Hemodialysis
MeSH Terms: conditions — Kidney Failure, Chronic; Renal Insufficiency; Renal Insufficiency, Chronic | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Intervention Model Description: A prospective, multi-center, single-arm study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Experimental: InnAVasc AVG treatment (Experimental): Patients will be surgically implanted with an InnAVasc Arteriovenous Graft (IG) in the forearm or upper arm using standard vascular surgical techniques. The graft will be placed in a "straight" (soft "C") configuration in the upper arm, or looped configuration in the forearm (forearm loop) or upper arm (axillary loop).
  Interventions: Device: InnAVasc Arteriovenous Graft (IG) surgical implant

INTERVENTIONS:
Device: InnAVasc Arteriovenous Graft (IG) surgical implant — The InnAVasc Arteriovenous Graft (IG) is a hemodialysis vascular access graft, intended for implantation in the lower or upper arm using standard vascular techniques, in patients requiring hemodialysis

SUMMARY:
The goal of the CSP-2002 clinical trial is to evaluate the safety and effectiveness of the InnAVasc Arteriovenous Graft (IG) for hemodialysis (HD) access in patients with end-stage renal disease (ESRD). The primary study endpoints are:

Primary Effectiveness Endpoint: The proportion of subjects with secondary patency at 6 months.

Primary Safety Endpoint: The incidence of device-related adverse events of special interest (AESIs) through 6 months.

Participants will be asked to sign an informed consent form. Once enrolled, they will be assessed to receive the study graft implant and asked to participate in periodic follow-up visits and assessments through 2 years following implant.

DETAILED DESCRIPTION:
The InnAVasc Arteriovenous Graft (IG) is intended for use in ESRD hemodialysis (HD) patients who require HD and whose next most appropriate access is an arteriovenous graft (AVG), also including those who may require an immediate cannulation AVG.

Patients with ESRD who require HD and are suitable for an AVG for HD access will be eligible for inclusion in the study. Subjects will be implanted with an InnAVasc Arteriovenous Graft (IG) in the forearm or upper arm using standard vascular surgical techniques. The graft will be placed in a "straight" (soft "C") configuration in the upper arm, or looped configuration in the forearm (forearm loop) or upper arm (axillary loop). Placing the graft across the elbow will be prohibited. Subjects must be able to be on antiplatelet therapy per the discretion of their physician (e.g., aspirin, clopidogrel, etc.).

ELIGIBILITY:
Inclusion Criteria:

Pre-Operative Inclusion Criteria:

Patients must meet the following criteria at screening in order to be scheduled for a procedure and potentially enrolled in the study:

1. Patients with ESRD whose next most appropriate option for AV access is placement of an AV graft to start or maintain hemodialysis therapy;
2. Age 18 to 90 years old, inclusive;
3. Suitable anatomy for implantation of upper arm "straight" or looped graft, or forearm looped graft (graft not to cross the bend of the elbow);
4. Ability to continue or commence antiplatelet therapy post graft implant (anticoagulation medication is acceptable if the subject is required to take an anticoagulant for a baseline medical condition);
5. Able and willing to give informed consent;
6. Anticipated life expectancy of at least 1 year.

Intra-Operative Inclusion Criteria:

Both vessels have been exposed and are deemed appropriate for implantation (i.e., based on the surgeon's opinion, artery is of adequate size, has adequate pulse to support AV access flow, is without significant calcification, and is safely clampable; and the vein is of adequate size, free of localized sclerosis, and is free of immediate outflow obstruction).

Pre-Operative Exclusion Criteria:

Patients will be excluded from the study at screening if they exhibit any of the following exclusion criteria:

1. History or evidence of severe cardiac disease (i.e., debilitating heart failure, or high risk of MI) in the opinion of the investigator which may preclude participation in and completion of the study;
2. Uncontrolled diabetes in the opinion of the investigator (i.e., multiple recent diabetes related hospitalizations);
3. For upper arm straight configuration, an antecubital fossa crease to axillary crease distance < 18 cm;
4. History or evidence of severe peripheral arterial disease in the extremity selected for implant (i.e., arterial inflow insufficient to support hemodialysis access);
5. Known or suspected central vein stenosis or obstruction on the side of planned graft implantation;
6. Baseline hypotension or history of frequent hypotensive episodes during dialysis that, in the opinion of the investigator, puts the patient at increased risk of graft thrombosis;
7. Uncontrolled hypertension, per the opinion of the investigator (i.e., recent history of recurrent hospitalizations for hypertensive related illness);
8. Baseline hemoglobin <7 g/dL;
9. Baseline platelet count <50,000 or >500,000 cells/mm3;
10. Documented history of stroke within 6 months prior to enrollment;
11. Treatment with any investigational drug or device within 30 days prior to enrollment;
12. Female patients who are pregnant, intending to become pregnant, nursing or intending to breastfeed during the study (pregnancy test may only be omitted, if patient is post-menopausal or has a documented history of hysterectomy or permanent sterilization);
13. History of cancer with active disease or treatment within the previous year, except for non-invasive basal or squamous cell carcinoma of the skin;
14. Immunodeficiency including documented history of human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS) or patients receiving immunosuppressive therapy for treatment of an acute inflammatory event or autoimmune flare. Chronic immunosuppressive therapy is acceptable;
15. Documented or suspected hypercoagulable condition;
16. Bleeding diathesis, other than that associated with ESRD;
17. Documented history of heparin-induced thrombocytopenia (HIT);
18. Active local or systemic infection as documented from the medical history or bloodwork/blood culture data. If the infection resolves, the subject must be at least one-week post resolution of that infection before implantation;
19. Scheduled renal transplant within 6 months;
20. Any other condition which in the judgment of the investigator would preclude adequate evaluation of the safety and effectiveness of the IG;
21. Patient is unable or unwilling to complete all required follow-up assessments and questionnaires.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Estimated)
Dates: Start 2020-12-03 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2029-07-01 (Estimated)

PRIMARY OUTCOMES:
Secondary patency of study device at 6 months | 6 months
  The primary effectiveness endpoint is defined as the proportion of subjects with secondary patency at 6 months.
Incidence of adverse events of special interest related to InnAVasc AVG [Time Frame: through 6 months] | 6 months
  The primary safety endpoint is the incidence of device-related adverse events of special interest (AESIs) through 6 months, defined as:
  1. Infection of the study graft;
  2. Pseudoaneurysm formation at any point along the study graft requiring surgical or endovascular intervention (pseudoaneurysms that occur at sites of needle cannulation, but which are small enough to be observed without intervention, do not trigger this element of the AESI endpoint);
  3. Bleeding from the study graft requiring surgical or endovascular intervention or ≥2-unit blood transfusion;
  4. Hematoma from the study graft requiring surgical or endovascular intervention;
  5. Seroma of the study graft requiring surgical or endovascular intervention;

SECONDARY OUTCOMES:
Successful cannulation on or before Postoperative Day 7 | 7 days
  Proportion of subjects achieving successful cannulation on or before Day 7, defined as the first 2-needle dialysis session through the study graft
Sustained use | 3, 6, 12, 18 and 24 months
  Proportion of subjects achieving sustained use of 3 months, 6, months, 12 months, 18 months and 24 months. Sustained use is a period of time in which the study graft is used for consecutive dialysis sessions without the requirement for alternative hemodialysis vascular access to be used as a route to receive renal replacement therapy. A sustained use period can be achieved at any time throughout the study period of 24 months.

OTHER OUTCOMES:
Primary Patency Rate | 3, 6, 12, 18 and 24 months
  Exploratory endpoint 1: Time from creation of access to first intervention to maintain patency or thrombosis
Assisted Primary Patency Rate | 3, 6, 12, 18 and 24 months
  Exploratory endpoint 2: Time from creation of access to first thrombosis, irrespective of intervention to maintain patency.
Secondary Patency Rate | 3, 6, 12, 18 and 24 months
  Exploratory endpoint 3: Time from creation of access to study graft abandonment or achievement of a censored event (death, transfer to peritoneal dialysis, renal transplant, steal, venous hypertension, or end of study period), and includes all surgical and endovascular interventions to reestablish study graft patency.
Thrombosis rate per patient | 3, 6, 12, 18 and 24 months
  Exploratory endpoint 4: The per patient rate of thrombosis events of the study graft at a particular timepoint.
Proportion of subjects achieving successful cannulation among those for whom it was attempted on or before Day 7 | First use of study graft
  Exploratory endpoint 5: Proportion of subjects achieving successful cannulation among those for whom it was attempted on or before Day 7, defined as the first 2-needle dialysis session through the study graft
Days of central venous catheter insitu | 3, 6, 12, 18 and 24 months
  Exploratory endpoint 6: Cumulative catheter days insitu
Incidence of individual adverse events | 3, 6, 12, 18 and 24 months
  Exploratory endpoint 7: cumulative adverse events, irrespective of device relatedness
Change from baseline Patient Reported Outcomes Measures/Patient Reported Experience Measures (PROM/PREM) survey (SF-VAQ); | 3, 6, 12, 18 and 24 months
  Exploratory endpoint 8: Change of responses over time from baseline
Intervention rate to restore or maintain patency | 3, 6, 12, 18 and 24 months
  Exploratory outcome 9: Intervention rate to restore or maintain patency (per patient per year)
Health Economics data analysis | 3, 6, 12, 18 and 24 months
  Exploratory endpoint 10: Health Economic data analysis to be performed based on available study data for the for treatment related costs (e.g. procedural costs, hospital costs, etc.)

CONTACTS AND LOCATIONS:
Overall Officials: John Ross, MD, Principal Investigator — MUSC Health Dialysis Access Institute
Locations (21):
- United States (21):
  - AKDHC Medical Research Services, LLC, Phoenix, Arizona
  - Sarasota Memorial Hospital, Sarasota, Florida
  - University of South Florida, Tampa, Florida
  - Piedmont Augusta, Augusta, Georgia
  - University of Louisville, Louisville, Kentucky
  - University of Maryland, Baltimore, Maryland
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Rutgers, Newark, New Jersey
  - Mount Sinai Hospital, New York, New York
  - Northwell Health, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Surgical Specialists of Charlotte, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - NC Heart and Vascular Research, LLC, Raleigh, North Carolina
  - WakeMed, Raleigh, North Carolina
  - Guthrie Clinic, Sayre, Pennsylvania
  - Prisma Health- Upstate, Greenville, South Carolina
  - Medical University of South Carolina, Orangeburg, South Carolina
  - Baylor Heart and Vascular, Dallas, Texas
  - Houston Methodist Hopsital, Houston, Texas
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gage SM, Lawson M, Nichols C, Sycks D, Manson RJ, Knight JA. An immediate access dialysis graft designed to prevent needle-related complications: Results from the initial pre-clinical studies. J Vasc Access. 2020 May;21(3):328-335. doi: 10.1177/1129729819874987. Epub 2019 Sep 16. PMID 31526086
- [Background] Gage SM, Illig KA, Ross JR. Use of a novel immediate access dialysis graft designed to prevent needle-related complications: A first-in-man case report. J Vasc Access. 2021 May;22(3):475-479. doi: 10.1177/1129729820917265. Epub 2020 May 5. PMID 32370648